CLINICAL TRIAL: NCT05309473
Title: Slow-wave Sleep Enhancement Using Acoustic Stimulation to Facilitate Performance Recovery During Restricted Sleep After Sleep Deprivation
Brief Title: Acoustic Stimulation During Restricted Sleep After Sleep Deprivation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, JOHN D. HUGHES, Neurologist, Walter Reed Army Institute of Research (WRAIR)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2901
Record Dates: First submitted 2022-02-17; First posted 2022-04-04 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Sleep Deprivation; Sleep Restriction; Acoustic Stimulation; Performance; Alertness
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Subjects Who Received Acoustic Stimulation (Experimental): Following 40 hours of deprivation participants will sleep for approximately a four hour recovery sleep period and receive acoustic stimulation via the Philips SmartSleep during slow-wave sleep. They will then sleep for second night of four hour recovery sleep and receive acoustic stimulation via the Philips Smart Sleep device during slow-wave sleep again.
  Interventions: Device: Philips SmartSleep Acoustic Stimulation Device
- Subjects Who Received Sham (no Acoustic Stimulation) (Sham Comparator): Following 40 hours of deprivation participants will sleep for approximately a four hour recovery sleep period and receive Sham (no acoustic stimulation) via the Philips SmartSleep during slow-wave sleep. They will then sleep for second night of four hour recovery sleep and receive Sham (no acoustic stimulation) via the Philips Smart Sleep device during slow-wave sleep again.
  Interventions: Device: Sham (no Acoustic Stimulation)

INTERVENTIONS:
Device: Philips SmartSleep Acoustic Stimulation Device — Prior to bedtime on the first two recovery nights, a Philips SmartSleep device will be applied to the head of each subject. Subjects will receive acoustic stimulation during the four hours of sleep.
  Arms: Subjects Who Received Acoustic Stimulation
Device: Sham (no Acoustic Stimulation) — Prior to bedtime on the first two recovery nights, a Philips SmartSleep device will be applied to the head of each subject. Subjects will receive Sham (no acoustic stimulation) during the four hours of sleep.
  Arms: Subjects Who Received Sham (no Acoustic Stimulation)

SUMMARY:
The purpose of this study is to determine if brief sounds or tones presented within a restricted period of recovery sleep after a period of sleep deprivation will enhance restorative properties and improve performance during a subsequent period of wakefulness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-pregnant, non-lactating women 18 to 39 years of age (inclusive)
* Must demonstrate adequate comprehension of the protocol, by achieving a score of at least 80% correct on a short multiple-choice quiz. Individuals who fail to achieve a passing score on the initial quiz will be given one opportunity to retest after a review of protocol information. Individuals who fail the comprehension assessment for the second time will be disqualified.

Exclusion Criteria:

* You must have learned English as your first language
* You must have a body mass index (BMI) below 30 (this is a mathematical calculation of your height and weight)
* You must not have current or a history of sleeping problems (for example, insomnia or sleep apnea), or symptoms that indicate a potential sleep disorder
* You must get an average of 6-9 hours of sleep per night and maintain a normal sleep/wake schedule
* You must not drink excessive amounts of caffeine, alcohol, or smoke cigarettes regularly
* You must not be on certain medications (determined on a case by case basis)
* You must test negative for illicit drugs
* Women must not be pregnant or nursing
* You must not be participating in another ongoing clinical trial
* You must have a social security number or tax identification number in order to be paid for screening and participation in the study
* You cannot have a history of the following conditions: Cardiovascular disease, a neurologic disorder, pulmonary disease requiring inhaler use, kidney disease or kidney abnormalities, liver disease of liver abnormalities, a history of psychiatric disorder requiring hospitalization or medication within the last two years or for a continuous period of more than 6 months in the last ten years

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Measure the effects of sleep deprivation/sleep restriction on performance using the Psychomotor Vigilance Task (PVT) | 8 days
  Performed at approximately 75 minutes intervals throughout the sleep deprivation and recovery days

SECONDARY OUTCOMES:
Measure simple arithmetic processing using the Mathematical Processing Subtest of the Automated Neuropsychological Assessment Metrics 4 (ANAM4) | 5 days
  Computer based series of mathematical calculations
Measure current mood states using the Mood Analogue Scale (MAS) | 5 days
  Computer based self adjective checklist of measure mood states
Measure latency to sleep using the Maintenance of Wakefulness Test (MWT) | 5 days
  Subjects will be escorted to their individual darkened, sound-attenuated bedrooms and allowed to lie down on their beds. They will be instructed to close their eyes and try to remain awake. Polysomnography will be monitored online.
Measure alertness using the Karolinska Sleepiness Scale (KSS) | 5 days
  Computer based self rated level of sleepiness
Measure various aspects of mood using the Walter Reed Army Institute of Research (WRAIR) Mood Battery | 5 days
  Computer based battery testing various aspects of mood
Measure various aspects of Sleep and Wakefulness using Polysomnographic measurements with video | 5 days
  Sleep will be measured during the night using polysomnography
Measure various aspects of Sleep and Wakefulness using Actigraphy | 22 days
  A watch-like device called an actigraph will measure movement to determine wake and sleep

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States